CLINICAL TRIAL: NCT05241574
Title: Radio(Chemo)Therapy Dose Escalation in Non-operative Management for Rectal Cancer: A Prospective NOM-3 Observational Study
Brief Title: Planned Non-operative Management for Rectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maria Sklodowska-Curie National Research Institute of Oncology (Other)
Responsible Party: Principal Investigator, Krzysztof Bujko, Clinical Professor, Maria Sklodowska-Curie National Research Institute of Oncology
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NOM-3
Record Dates: First submitted 2022-01-25; First posted 2022-02-15 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Rectal Cancer
Keywords: Rectal cancer; Non-operative management
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Intervention Model Description: A dose escalation study, either radiotherapy dose escalation or chemotherapy dose escalation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- radiotherapy dose escalation (Experimental): Additional two fractions of endorectal high dose rate iridium brachytherapy boost, 10 Gy each.
  Interventions: Radiation: Radiotherapy boost
- chemotherapy dose escalation (Experimental): Additional three cycles of consolidation chemotherapy consisted of 5-fluorouracil, leucovorin and oxaliplatin (FOLFOX4).
  Interventions: Drug: Additional consolidation chemotherapy

INTERVENTIONS:
Radiation: Radiotherapy boost — Additional endorectal high rate irydium brachytherapy boost, 2 fractions of 10 Gy each.
  Arms: radiotherapy dose escalation
Drug: Additional consolidation chemotherapy — Three additional cycles of 5-fluorouracil, leucovorin and oxaliplatin (FOLFOX4) consolidation chemotherapy
  Arms: chemotherapy dose escalation

SUMMARY:
The investigators propose to conduct an observational study on consecutive patients with low-lying or mid rectal cancers smaller than 5 cm in length and less than 50% of rectal circumferential extent. The aim of this study is to test a hypothesis that escalation of either radiation or chemotherapy dose of the routine preoperative radio(chemo)therapy leads to an increase of clinical complete response rate. The planned sample size of 23 patients was calculated based on the assumption that clinical complete response rate after routine preoperative radio(chemo)therapy is 34% [1] and expected rate after radio(chemo)therapy dose escalation is 75% [2-4]. An endorectal high dose rate iridium brachytherapy boost (2 fractions of 10 Gy) will be added after the routine preoperative treatment consisted of external beam radiotherapy (5 × 5 Gy) combined with sequential 3 cycles of consolidation FOLFOX4. However, for patients with involvement of the anal canal, additional 3 cycles of consolidation FOLFOX4 (6 cycles in total) will be added instead of brachytherapy boost to avoid severe post-radiation toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Adenocarcinoma of the rectum classified clinically as T2, T3a-c or T4b but only with superficial infiltration of the vagina or prostate; tumour accessible by digital rectal examination; tumour ≤5 cm in length and ≤50% of rectal circumferential extent; N0-N2, but mesorectal node <7 mm and no lateral nodes enlargement); extramural vascular invasion but not larger than 7 mm in the largest dimension; M0.
2. Operable patient
3. Patient having read the information note and having signed the informed consent
4. Follow-up possible

Exclusion Criteria:

1. Inoperable patient
2. cT1, cT3d, large T4, tumour ≥5cm or ≥50 of rectal circumferential extent
3. Enlargement of lateral nodes or any node ≥8 mm in diameter
4. Patient presenting metastasis at diagnosis
5. Previous pelvic irradiation
6. Simultaneous progressive another cancer
7. Close follow-up uncertain.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2021-08-03 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Rate of patients with clinical complete response. | 15 weeks from the radiation start
  Clinical complete response will be assessed by digital rectal examination, endoscopy and MRI. The analysis will take place 6 months after the start of treatment of a last enrolled patient.

SECONDARY OUTCOMES:
Regrowth rate. | From 12 months to 26 months from the radiation start.
  Regrowth rate will be accessed at 2 years in patients undergoing watch-and-wait. The analysis will take place 12 months after the start of treatment of a last enrolled patient.
Anorectal function. | One year after the radiation start.
  Anorectal function will be assessed by LARS scale before treatment and one year after the radiation start.
Acute and late toxicity assessed by Common Terminology Criteria for Adverse Events (CTCAE), version 5. | From 12 months to 26 months from the radiation start.
  Acute and late toxicity will be assessed by CTCAE v.5 scale.

CONTACTS AND LOCATIONS:
Overall Officials: Paulina Śliwka, MS, Study Director — Maria Skłodowska-Curie National Research Institute of Oncology
Locations (1):
- M. Skłodowska-Curie National Research Institute of Oncology, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Jankowski M, Pietrzak L, Rupinski M, Michalski W, Holdakowska A, Paciorek K, Rutkowski A, Olesinski T, Cencelewicz A, Szczepkowski M, Zegarski W, Reszke J, Richter P, Wawok P, Malecki K, Bebenek M, Szelachowska J, Mazurek M, Gisterek I, Polkowski W, Jankiewicz M, Stylinski R, Socha J, Bujko K; Polish Colorectal Study Group. Watch-and-wait strategy in rectal cancer: Is there a tumour size limit? Results from two pooled prospective studies. Radiother Oncol. 2021 Jul;160:229-235. doi: 10.1016/j.radonc.2021.05.014. Epub 2021 May 21. PMID 34023328
- [Background] Garant A, Magnan S, Devic S, Martin AG, Boutros M, Vasilevsky CA, Ferland S, Bujold A, DesGroseilliers S, Sebajang H, Richard C, Vuong T. Image Guided Adaptive Endorectal Brachytherapy in the Nonoperative Management of Patients With Rectal Cancer. Int J Radiat Oncol Biol Phys. 2019 Dec 1;105(5):1005-1011. doi: 10.1016/j.ijrobp.2019.08.042. Epub 2019 Aug 30. PMID 31476417
- [Background] Rijkmans EC, Cats A, Nout RA, van den Bongard DHJG, Ketelaars M, Buijsen J, Rozema T, Franssen JH, Velema LA, van Triest B, Marijnen CAM. Endorectal Brachytherapy Boost After External Beam Radiation Therapy in Elderly or Medically Inoperable Patients With Rectal Cancer: Primary Outcomes of the Phase 1 HERBERT Study. Int J Radiat Oncol Biol Phys. 2017 Jul 15;98(4):908-917. doi: 10.1016/j.ijrobp.2017.01.033. Epub 2017 Jan 20. PMID 28366579
- [Background] 4. Garcia-Aguilar J, Patil S, Kim JK, et al. Preliminary results of the organ preservation of rectal adenocarcinoma (OPRA) trial. J Clin Oncol 38: 2020 (suppl; abstr 4008).